CLINICAL TRIAL: NCT04404816
Title: Effects of Non-invasive Ventilation With Helium-oxygen Mixture in Premature Infants With Respiratory Distress Syndrome on Pulmonary Function and Electric Activity of the Diaphragm
Brief Title: Effects of Non-invasive Ventilation With Helium-oxygen Mixture in Premature Infants With Respiratory Distress Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: European Society for Paediatric Research (Unknown)
Responsible Party: Principal Investigator, Tomasz Szczapa, Deputy Head - Department of Neonatology; Head - Neonatal Biophysical Monitoring and Cardiopulmonary Therapies Research Unit, Poznan University of Medical Sciences
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 072015
Record Dates: First submitted 2020-05-05; First posted 2020-05-28 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Distress Syndrome; Premature Infants
Keywords: heliox; respiratory distress syndrome (RDS); non-invasive ventilation; NIRS; EaDI; Edi; NIV; NAVA; helium-oxygen
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — heliox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): premature infants born < 33 G.A. enrolled in the first 72 hours after birth, with respiratory distress syndrome, requiring non-invasive ventilation with FiO2 <0.4
  Interventions: Drug: heliox
- Group 2 (Experimental): premature infants born < 33 G.A. with respiratory insufficiency requiring mechanical ventilation, after more than 1 failed extubation attempt
  Interventions: Drug: heliox

INTERVENTIONS:
Drug: heliox — NIV-NAVA with a conventional gas mixture (air-oxygen) at baseline, 3 hours of NIV-NAVA with heliox and return to NIV-NAVA with air-oxygen.
  Other Names: helium-oxygen gas mixture

SUMMARY:
The use of a mixture of helium with oxygen (heliox) as a breathing gas may be beneficial due to its unique physical properties, such as low density and high carbon dioxide (CO2) diffusion coefficient. In previous studies in neonates with respiratory failure, conventional ventilation with heliox was associated with improved oxygenation and selected respiratory parameters. The use of heliox may increase the effectiveness of intermittent nasal positive pressure ventilation (NIPPV), but knowledge about the effects of such therapy on newborns is limited.The use of non- invasive neurally adjusted ventilatory assist (NIV-NAVA) allows synchronization and assessment of electrical activity of the diaphragm (EaDI) during heliox administration in premature babies with respiratory failure.

DETAILED DESCRIPTION:
Aim of the study was to assess of the impact of non-invasive ventilation with heliox on respiratory function, diaphragm bioelectrical activity, cerebral oxygenation and selected vital signs in premature neonates with respiratory failure. 23 neonates ≤32 weeks gestational age (GA) were enrolled in the study. Patients were eligible for inclusion when ventilated due to respiratory failure, and in group 1 (n=12) on NIV as primary modality with oxygen requirement of 0.25-0.4 in the first 72 hours of life, or in group 2 (n=11) ready to extubate according to the given criteria. Newborns were ventilated with NIV NAVA and standard breathing gas (air-oxygen) at baseline. Heliox was introduced for 3 hours, followed by 3 hours of air-oxygen. NAVA level was kept constant and pulse oximeter oxygen saturation (SpO2) kept in range of 90-95%. Recorded parameters included heart rate (HR), SpO2 and cerebral tissue oxygenation (StO2). Selected ventilation parameters: peak inspiratory pressure (PIP), positive end-expiratory pressure (PEEP), mean airway pressure (MAP), air leakage during NIV, fraction of inspired oxygen (FiO2) as well as electrical activity of the diaphragm (EaDI mean, minimum and maximum) were also acquired. Blood gas analysis was performed in each period of the study. Statistical analysis was completed with ANOVA Friedman's test and single-factor repeated-measures analysis of variance.

ELIGIBILITY:
Inclusion Criteria (Group 1):

* GA under 33 weeks GA
* Need for NIV due to clinical symptoms of respiratory distress in course of RDS
* FiO2=0.25-0.4
* Enrollment within first 72 hours of life
* Parental consent

Inclusion Criteria (Group 2):

* GA under 33 weeks GA
* Need for MV due to clinical symptoms of respiratory distress
* at least one failed attempted extubation
* Parental consent

Exclusion Criteria:

* Major congenital anomalies
* Deteriorating pulmonary function despite NIV and the need for intubation and conventional mechanical ventilation (CMV) (Preliminary criteria: pH< 7.22, carbon dioxide partial pressure (pCO2) >65)

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
baseline minimal electric activity of the diaphragm (EaDI min) | measured at baseline
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV, microvolts] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
baseline mean electric activity of the diaphragm (EaDI mean) | measured at baseline
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
baseline maximal electric activity of the diaphragm (EaDI max) | measured at baseline
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
minimal electric activity of the diaphragm (EaDI min) after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
mean electric activity of the diaphragm (EaDI mean) after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
maximal electric activity of the diaphragm (EaDI max) after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
minimal electric activity of the diaphragm (EaDI min) after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
mean electric activity of the diaphragm (EaDI mean) after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
maximal electric activity of the diaphragm (EaDI max) after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
minimal electric activity of the diaphragm (EaDI min) after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
mean electric activity of the diaphragm (EaDI mean) after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
maximal electric activity of the diaphragm (EaDI max) after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
minimal electric activity of the diaphragm (EaDI min) after 15 minutes of standard mixture | measured after 15 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
mean electric activity of the diaphragm (EaDI mean) after 15 minutes of standard mixture | measured after 15 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
maximal electric activity of the diaphragm (EaDI max) after 15 minutes of standard mixture | measured after 15 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
minimal electric activity of the diaphragm (EaDI min) after 60 minutes of standard mixture | measured after 60 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
mean electric activity of the diaphragm (EaDI mean) after 60 minutes of standard mixture | measured after 60 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
maximal electric activity of the diaphragm (EaDI max) after 60 minutes of standard mixture | measured after 60 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
minimal electric activity of the diaphragm (EaDI min) after 180 minutes of standard mixture | measured after 180 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI min [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
mean electric activity of the diaphragm (EaDI mean) after 180 minutes of standard mixture | measured after 180 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI mean [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
maximal electric activity of the diaphragm (EaDI max) after 180 minutes of standard mixture | measured after 180 minutes since the return to ventilation with standard mixture
  Using the NAVA (neurally adjusted ventilatory assist) module of the Maquet Servo-i ventilator and "Servo-tracker" software EaDI max [mcV] values will be recorded during the study and their values will be compared between the heliox and air-oxygen NIV (non -invasive ventilation).
baseline PIP (peak inspiratory pressure) | measured at baseline
  PIP [cm H2O, centimeters of water] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
baseline PEEP (positive end-expiratory pressure) | measured at baseline
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
baseline MAP (mean airway pressure) | measured at baseline
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PIP (peak inspiratory pressure) after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  PIP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PIP (peak inspiratory pressure) after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  PIP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PIP (peak inspiratory pressure) after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  PIP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PIP (peak inspiratory pressure) after 15 minutes of standard mixture | measured after 15 minutes since the return to ventilation with standard mixture
  PIP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PIP (peak inspiratory pressure) after 60 minutes of standard mixture | measured after 60 minutes since the return to ventilation with standard mixture
  PIP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PIP (peak inspiratory pressure) after 180 minutes of standard mixture | measured after 180 minutes since the return to ventilation with standard mixture
  PIP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PEEP (positive end-expiratory pressure) after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PEEP (positive end-expiratory pressure) after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PEEP (positive end-expiratory pressure) after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PEEP (positive end-expiratory pressure) after 15 minutes of standard mixture | measured after 15 minutes since the return to ventilation with standard mixture
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PEEP (positive end-expiratory pressure) after 60 minutes of standard mixture | measured after 60 minutes since the return to ventilation with standard mixture
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
PEEP (positive end-expiratory pressure) after 180 minutes of standard mixture | measured after 180 minutes since the return to ventilation with standard mixture
  PEEP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
MAP (mean airway pressure) after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
MAP (mean airway pressure) after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
MAP (mean airway pressure) after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
MAP (mean airway pressure) after 15 minutes of standard ventilation | measured after 180 minutes since the return to ventilation with standard mixture
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
MAP (mean airway pressure) after 60 minutes of standard ventilation | measured after 60 minutes since the return to ventilation with standard mixture
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
MAP (mean airway pressure) after 180 minutes of standard ventilation | measured after 180 minutes since the return to ventilation with standard mixture
  MAP [cm of water / cm H2O] will be recorded by Servo-tracker software and the values will be compared between the heliox and air-oxygen NIV.
baseline NIV leakage | measured at baseline
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.
NIV leakage after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.
NIV leakage after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.
NIV leakage after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.
NIV leakage after 15 minutes of standard mixture | measured after 15 minutes since the return to ventilation with standard mixture
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.
NIV leakage after 60 minutes of standard mixture | measured after 60 minutes since the return to ventilation with standard mixture
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.
NIV leakage after 180 minutes of standard mixture | measured after 180 minutes since the return to ventilation with standard mixture
  gas leakage fraction [%] during NIV (non-invasive ventilation) recorded by Servo-tracker software their values will be compared between the heliox and air-oxygen NIV.

SECONDARY OUTCOMES:
baseline cerebral oxygenation | measured at baseline
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
Cerebral oxygenation after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
Cerebral oxygenation after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
Cerebral oxygenation after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
Cerebral oxygenation after 15 minutes of standard mixture | measured after 15 minutes since the return to standard mixture ventilation
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
Cerebral oxygenation after 60 minutes of standard mixture | measured after 60 minutes since the return to standard mixture ventilation
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
Cerebral oxygenation after 180 minutes of standard mixture | measured after 180 minutes since the return to standard mixture ventilation
  Cerebral tissue oxygen saturation (StO2; [%]) measured with near infrared spectroscopy (NIRS) - NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA - their values will be compared between the heliox and air-oxygen NIV.
baseline oxygen requirements | recorded at baseline
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
oxygen requirements after 15 minutes of heliox | recorded after 15 minutes of heliox ventilation
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
oxygen requirements after 60 minutes of heliox | recorded after 60 minutes of heliox ventilation
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
oxygen requirements after 180 minutes of heliox | recorded after 180 minutes of heliox ventilation
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
oxygen requirements after 15 minutes of standard ventilation | recorded after 15 minutes since the return to standard mixture ventilation
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
oxygen requirements after 60 minutes of standard ventilation | recorded after 60 minutes since the return to standard mixture ventilation
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
oxygen requirements after 180 minutes of standard ventilation | recorded after 180 minutes since the return to standard mixture ventilation
  Fraction of inspired oxygen (FiO2) will be recorded during heliox and air-oxygen NIV to maintain the saturation assessed by pulse oximetry (SpO2) in 90-95% range; their values will be compared between the phases of the study
baseline capillary blood gas analysis | blood samples drawn at baseline
  Cobas B 221; Roche, Germany; the values will be compared between the heliox and air-oxygen NIV.
capillary blood gas analysis after 3 hours of heliox | blood samples drawn after 3 hours of heliox ventilation
  Cobas B 221; Roche, Germany; the values will be compared between the heliox and air-oxygen NIV.
capillary blood gas analysis after 3 hours of standard mixture | blood samples drawn after 3 hours of standard mixture ventilation
  Cobas B 221; Roche, Germany; the values will be compared between the heliox and air-oxygen NIV.
baseline heart rate | measured at baseline
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
heart rate after 15 minutes of heliox | measured after 15 minutes of heliox ventilation
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
heart rate after 60 minutes of heliox | measured after 60 minutes of heliox ventilation
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
heart rate after 180 minutes of heliox | measured after 180 minutes of heliox ventilation
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
heart rate after 15 minutes of standard mixture | measured after 15 minutes since the return to standard mixture ventilation
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
heart rate after 60 minutes of standard mixture | measured after 60 minutes since the return to standard mixture ventilation
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
heart rate after 180 minutes of standard mixture | measured after 180 minutes since the return to standard mixture ventilation
  heart rate (HR, [bpm / beats per minute]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA), values will be compared between the heliox and air-oxygen NIV.
baseline oxygen saturation | measured at baseline
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.
oxygen saturation after 15 minutes of heliox | measured 15 minutes after heliox ventilation
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.
oxygen saturation after 60 minutes of heliox | measured 60 minutes after heliox ventilation
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.
oxygen saturation after 180 minutes of heliox | measured 180 minutes after heliox ventilation
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.
oxygen saturation after 15 minutes of standard mixture | measured 15 minutes since the return to standard mixture ventilation
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.
oxygen saturation after 60 minutes of standard mixture | measured 60 minutes since the return to standard mixture ventilation
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.
oxygen saturation after 180 minutes of standard mixture | measured 180 minutes since the return to standard mixture ventilation
  SpO2 (peripheral capillary oxygen saturation, [%]) measured by NONIN Sen Smart Model X-100, Nonin Medical Inc., Plymouth, USA) and the values will be compared between the heliox and air-oxygen NIV.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Szczapa, M.D. PhD, Study Director — Department of Neonatology - Poznan University of Medical Sciences
Locations (1):
- Gynecological and obstetric teaching hospital, Departament of Neonatology, Polna street 33, Poznan, Great Poland, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Halliday HL; European Association of Perinatal Medicine. European consensus guidelines on the management of neonatal respiratory distress syndrome in preterm infants--2013 update. Neonatology. 2013;103(4):353-68. doi: 10.1159/000349928. Epub 2013 May 31. PMID 23736015
- [Background] Elleau C, Galperine RI, Guenard H, Demarquez JL. Helium-oxygen mixture in respiratory distress syndrome: a double-blind study. J Pediatr. 1993 Jan;122(1):132-6. doi: 10.1016/s0022-3476(05)83506-1. PMID 8419600
- [Background] Colnaghi M, Pierro M, Migliori C, Ciralli F, Matassa PG, Vendettuoli V, Mercadante D, Consonni D, Mosca F. Nasal continuous positive airway pressure with heliox in preterm infants with respiratory distress syndrome. Pediatrics. 2012 Feb;129(2):e333-8. doi: 10.1542/peds.2011-0532. Epub 2012 Jan 30. PMID 22291116
- [Background] Szczapa T, Gadzinowski J, Moczko J, Merritt TA. Heliox for mechanically ventilated newborns with bronchopulmonary dysplasia. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F128-33. doi: 10.1136/archdischild-2013-303988. Epub 2013 Nov 15. PMID 24239984
- [Background] Szczapa T, Gadzinowski J. Use of heliox in the management of neonates with meconium aspiration syndrome. Neonatology. 2011;100(3):265-70. doi: 10.1159/000327531. Epub 2011 Jun 23. PMID 21701217
- [Background] Jassar RK, Vellanki H, Zhu Y, Hesek A, Wang J, Rodriguez E, Wu J, Shaffer TH, Wolfson MR. High flow nasal cannula (HFNC) with Heliox decreases diaphragmatic injury in a newborn porcine lung injury model. Pediatr Pulmonol. 2014 Dec;49(12):1214-22. doi: 10.1002/ppul.23000. Epub 2014 Feb 5. PMID 24500982
- [Background] Sinderby C, Beck J, Spahija J, Weinberg J, Grassino A. Voluntary activation of the human diaphragm in health and disease. J Appl Physiol (1985). 1998 Dec;85(6):2146-58. doi: 10.1152/jappl.1998.85.6.2146. PMID 9843538
- [Background] Beck J, Reilly M, Grasselli G, Qui H, Slutsky AS, Dunn MS, Sinderby CA. Characterization of neural breathing pattern in spontaneously breathing preterm infants. Pediatr Res. 2011 Dec;70(6):607-13. doi: 10.1203/PDR.0b013e318232100e. PMID 21857389
- [Background] Brooks LJ, DiFiore JM, Martin RJ. Assessment of tidal volume over time in preterm infants using respiratory inductance plethysmography, The CHIME Study Group. Collaborative Home Infant Monitoring Evaluation. Pediatr Pulmonol. 1997 Jun;23(6):429-33. doi: 10.1002/(sici)1099-0496(199706)23:63.0.co;2-d. PMID 9220525
- [Background] Nawab US, Touch SM, Irwin-Sherman T, Blackson TJ, Greenspan JS, Zhu G, Shaffer TH, Wolfson MR. Heliox attenuates lung inflammation and structural alterations in acute lung injury. Pediatr Pulmonol. 2005 Dec;40(6):524-32. doi: 10.1002/ppul.20304. PMID 16193495
- [Background] Kuligowski J, Escobar J, Quintas G, Lliso I, Torres-Cuevas I, Nunez A, Cubells E, Rook D, van Goudoever JB, Vento M. Analysis of lipid peroxidation biomarkers in extremely low gestational age neonate urines by UPLC-MS/MS. Anal Bioanal Chem. 2014 Jul;406(18):4345-56. doi: 10.1007/s00216-014-7824-6. Epub 2014 May 11. PMID 24817352
- [Background] Kuligowski J, Torres-Cuevas I, Quintas G, Rook D, van Goudoever JB, Cubells E, Asensi M, Lliso I, Nunez A, Vento M, Escobar J. Assessment of oxidative damage to proteins and DNA in urine of newborn infants by a validated UPLC-MS/MS approach. PLoS One. 2014 Apr 2;9(4):e93703. doi: 10.1371/journal.pone.0093703. eCollection 2014. PMID 24695409
- [Background] Oei GT, Weber NC, Hollmann MW, Preckel B. Cellular effects of helium in different organs. Anesthesiology. 2010 Jun;112(6):1503-10. doi: 10.1097/ALN.0b013e3181d9cb5e. PMID 20460992